CLINICAL TRIAL: NCT02382666
Title: A Phase 1, 2-Part, Single Ascending Dose Assessment of the Safety, Tolerability, and Pharmacokinetics of Rolapitant Intravenous in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-11-5022-C
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — rolapitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rolapitant Cohort 1 (Experimental): Investigational Product: Rolapitant Dose 1 administered IV as a 30-minute infusion Dosage Form: 2 mg/mL solution
  Interventions: Drug: Rolapitant
- Rolapitant Cohort 2 (Experimental): Investigational Product: Rolapitant Dose 2 administered IV as a 30-minute infusion Dosage Form: 2 mg/mL solution
  Interventions: Drug: Rolapitant
- Rolapitant Cohort 3 (Experimental): Investigational Product: Rolapitant Dose 3 administered IV as a 30-minute infusion Dosage Form: 2 mg/mL solution
  Interventions: Drug: Rolapitant
- Rolapitant Cohort 4 (Experimental): Investigational Product: Rolapitant Dose 4 administered IV as a 30-minute infusion Dosage Form: 2 mg/mL solution
  Interventions: Drug: Rolapitant
- Rolapitant Cohort 5 (Experimental): Investigational Product: Rolapitant Dose 5 administered IV as a 30-minute infusion Dosage Form: 2 mg/mL solution
  Interventions: Drug: Rolapitant
- Rolapitant Cohort 6 (Experimental): Investigational Product: Rolapitant Dose 6 administered IV as a 30-minute infusion Dosage Form: 2 mg/mL solution
  Interventions: Drug: Rolapitant

INTERVENTIONS:
Drug: Rolapitant

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single increasing doses of intravenously administered rolapitant in healthy male and female subjects.

DETAILED DESCRIPTION:
Part 1 of the study is designed to evaluate the safety and tolerability of a SAD, up to 6 cohorts,of rolapitant IV (2 mg/mL solution) administered as an IV infusion over 30 minutes.

In Part 2 of the study, the safety and tolerability of the highest safe and well-tolerated dose established in Part 1 will be evaluated in an expanded cohort. The highest safe and well-tolerated dose established in Part 1 will be ascertained by the following criteria: an upper limit of 90% confidence interval (CI) for Cmax. A minimum of 40 subjects will be enrolled in Part 2.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject must be a healthy male or female aged 18 to 55 years at Screening
* A female subject must have a negative pregnancy test at Screening and on Day -1.
* A female subject of childbearing potential must agree to use an accepted method of birth control (excluding hormonal birth control methods) from Screening through 30 days after final study drug administration.
* Subject must have a body mass index (BMI) from 18.5 to 32.0 kg/m2 and a weight of

  ≥ 50 kg at Screening.
* Subject must be able to provide informed consent after risks and benefits have been explained. Subject must also be willing and able to comply with the protocol requirements.
* Subject must be in general good health as determined by the Investigator based on pre-study medical, medication, and surgical history; physical examination; and clinical laboratory tests.

Main Exclusion Criteria:

* Subject must not have been dosed with test drug or blinded study drug in another investigational study within 30 days or 5 half-lives of the biologic activity of the test drug, whichever is longer, before the time of first study dose.
* Subject must not have a history of hypersensitivity to rolapitant IV or any of its excipients or who have completed a study visit as part of a previous rolapitant study within the 6 months prior to first study drug administration (Day
* Subject must not have poor venous access or consider venipuncture intolerable.
* Subject must not have a history of significant complications or anxiety associated with the IV administration of medications that, in the opinion of the Investigator, could make the subject unable to complete dosing requirements.
* Subject must not be pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Part 1 Dose Escalation: Safety and Tolerability (adverse events) | 0-30 days after administration of study drug
  To evaluate the safety and tolerability of rolapitant IV (30 minutes infusion) in healthy adult volunteers as assessed by the incidence and severity of AEs
Part 2 Dose Treatment: Safety and Tolerability (adverse events) | : 0-30 days after administration of study drug
  To evaluate the safety and tolerability of rolapitant IV (30 minutes infusion) to an expanded cohort of healthy adult volunteers at the highest safe and well-tolerated dose established in Part 1 as assessed by the incidence and severity of AEs.

SECONDARY OUTCOMES:
1. AUC0-last: area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration | 0-21 days
2. Cmax = observed maximum plasma concentration | 0-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vargo, MD, Study Director — Tesaro, Inc.
Locations (1):
- Parexel, Baltimore, Maryland, United States